CLINICAL TRIAL: NCT01614964
Title: Phase 2 Proof of Concept Study of a Candidate Aminoquinoline Antimalarial (AQ-13)
Brief Title: Studies of a Candidate Aminoquinoline Antimalarial (AQ-13)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Tulane University (Other)
Collaborators: University of the Sciences, Techniques and Technologies of Bamako (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2149; FDA 1R01-FD-003373 (Other Grant/Funding Number: FDA Office of Orphan Products Development)
Record Dates: First submitted 2012-06-06; First posted 2012-06-08 (Estimated); Results first posted 2024-07-11 (Actual); Last update posted 2024-07-11 (Actual); Status verified 2024-06

CONDITIONS: Malaria
Keywords: Plasmodium falciparum; pharmacokinetics; antimalarials (antimalarial drugs); chloroquine (chloroquine-resistant); QT (QTc) interval
MeSH Terms: conditions — Malaria; Malaria, Falciparum

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- AQ-13 (Experimental): Adult Malian males 18 years of age or older with uncomplicated P. falciparum malaria who agree to participate and provide their informed consent will be randomized to receive treatment with either AQ-13 or Coartem. Intervention 'AQ-13 Treatment' Participants randomized to the AQ-13 arm will be treated with two (350 mg) capsules on days 1 and 2 and one (350 mg) AQ-13 capsule on day 3 for a total oral dose of 1750 mg of AQ-13 (5 capsules containing 350 mg apiece) over 3 days.
  Interventions: Drug: AQ-13 Treatment
- Coartem Treatment (Active Comparator): Adult Malian males 18 years of age or older with uncomplicated P. falciparum malaria who agree to participate and provide their informed consent will be randomized to receive treatment with either AQ-13 or Coartem. Intervention: Active Comparator: Coartem. Participants randomized to the Coartem arm will be treated with 80 mg artemether and 480 mg lumefantrine at the time of diagnosis and 8 hours later on day 1, the same doses (80 mg artemether and 480 mg lumefantrine) twice on day 2 (24 and 36 hours after diagnosis) and twice more on day 3 (48 and 60 hours after diagnosis) for total oral doses of 480 mg artemether and 2880 mg lumefantrine over 3 days.
  Interventions: Drug: Coartem Treatment

INTERVENTIONS:
Drug: AQ-13 Treatment — Adult Malian males 18 years of age or older with uncomplicated P. falciparum malaria who agree to participate and provide their informed consent will be randomized to receive treatment with either AQ-13 or Coartem. Intervention 'AQ-13 Treatment' Participants randomized to the AQ-13 arm will be treated with two (350 mg) capsules on days 1 and 2 and one (350 mg) AQ-13 capsule on day 3 for a total oral dose of 1750 mg of AQ-13 (5 capsules containing 350 mg apiece) over 3 days.
  Other Names: N'-(7-Chloroquinolin-4-yl)-N,N-diethyl-propane-1,3-diamine.
  Arms: AQ-13
Drug: Coartem Treatment — Adult Malian males 18 years of age or older with uncomplicated P. falciparum malaria who agree to participate and provide their informed consent will be randomized to receive treatment with either AQ-13 or Coartem. Intervention 'Coartem Treatment' Participants randomized to the Coartem arm will receive six doses of Coartem tablets over 3 days (each dose containing 80 mg artemether and 480 mg lumefantrine). Those six doses will be given at the time of diagnosis and 8 hours later on day 1, at 24 and 36 hours on day 2 and at 48 and 60 hours on day 3 for total doses of 480 mg artemether and 2880 mg lumefantrine over 3 days.
  Other Names: Tablets contain 20 (or 80) mg artemether and 120 (or 480) mg lumefantrine.
  Arms: Coartem Treatment

SUMMARY:
This is an initial efficacy study of a candidate antimalarial in human subjects with uncomplicated malaria caused by the most common and most important parasite in Africa (Plasmodium falciparum). This study will enroll 66 adult Malian males with uncomplicated P. falciparum malaria and randomize them to treatment with 1750 mg of the investigational drug (AQ-13) by mouth over 3 days or the current standard treatment, which is 2 doses of Coartem twice daily for 3 days. The hypothesis underlying this study is that AQ-13 will be similarly effective to Coartem for the treatment of uncomplicated P. falciparum malaria due to both chloroquine-susceptible and chloroquine-resistant parasites. Funding Source - FDA Office of Orphan Product Development (OOPD).

DETAILED DESCRIPTION:
This is an initial efficacy study (Phase 2 Proof of Concept Study) of a candidate antimalarial in human subjects with uncomplicated malaria caused by the most common and most important parasite in Africa (Plasmodium falciparum). This study will enroll 66 adult Malian males with uncomplicated P. falciparum malaria and randomize them to treatment with 1750 mg of the investigational drug (AQ-13) by mouth over 3 days or the current standard treatment, which is 80 mg of artemether and 480 mg of lumefantrine twice daily for 3 days. The hypothesis underlying this study is that AQ-13 will be similarly effective to Coartem for the treatment of uncomplicated P. falciparum malaria due to both chloroquine-susceptible and chloroquine-resistant parasites.

ELIGIBILITY:
Inclusion Criteria

1. Adult Malian males ≥ 18 years of age,
2. Uncomplicated malaria with ≥ 2,000 asexual P. falciparum parasites per ul, and
3. Informed consent obtained and signed.

Exclusion Criteria

1. Severe or complicated malaria (including temperature ≥ 40o C),
2. ≥ 100,000 asexual parasites per ul of blood,
3. Anemia or other laboratory results (other than malaria) that require treatment (e.g., Hb ≤ 7 gm/dL, K+ ≤ 3.5 millimolar (mM), BP ≥ 140/90),
4. Seizures or impaired consciousness,
5. Recent antimalarial treatment by history (within ≤ 2 weeks),
6. Chronic medications (including inducers of Cytochrome P450 3A4 [CYP3A4] activity such as rifampin and nevirapine),
7. Ventricular or atrial arrhythmias, or second or third degree heart block on the screening ECG or Holter recording,
8. Infection with other plasmodial species on the blood smear (P. ovale, P. ovale, P. vivax).

Ages: 18 Years to 99 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2013-08 (Actual); Primary Completion 2016-01 (Actual); Study Completion 2017-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Donald J. Krogstad, MD, Principal Investigator — Tulane School of Public Health and Tropical Medicine
Locations (1):
- Clinical Research Center (Hopital Point G, University of the Sciences, Techniques and Technologies of Bamako), Bamako, Mali

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] De D, Krogstad FM, Cogswell FB, Krogstad DJ. Aminoquinolines that circumvent resistance in Plasmodium falciparum in vitro. Am J Trop Med Hyg. 1996 Dec;55(6):579-83. doi: 10.4269/ajtmh.1996.55.579. PMID 9025680
- [Background] De D, Krogstad FM, Byers LD, Krogstad DJ. Structure-activity relationships for antiplasmodial activity among 7-substituted 4-aminoquinolines. J Med Chem. 1998 Dec 3;41(25):4918-26. doi: 10.1021/jm980146x. PMID 9836608
- [Background] Ramanathan-Girish S, Catz P, Creek MR, Wu B, Thomas D, Krogstad DJ, De D, Mirsalis JC, Green CE. Pharmacokinetics of the antimalarial drug, AQ-13, in rats and cynomolgus macaques. Int J Toxicol. 2004 May-Jun;23(3):179-89. doi: 10.1080/10915810490471352. PMID 15204721
- [Background] Deng H, Liu H, Krogstad FM, Krogstad DJ. Sensitive fluorescence HPLC assay for AQ-13, a candidate aminoquinoline antimalarial, that also detects chloroquine and N-dealkylated metabolites. J Chromatogr B Analyt Technol Biomed Life Sci. 2006 Apr 3;833(2):122-8. doi: 10.1016/j.jchromb.2005.12.011. Epub 2006 Jan 18. PMID 16520100
- [Background] Hocart SJ, Liu H, Deng H, De D, Krogstad FM, Krogstad DJ. 4-aminoquinolines active against chloroquine-resistant Plasmodium falciparum: basis of antiparasite activity and quantitative structure-activity relationship analyses. Antimicrob Agents Chemother. 2011 May;55(5):2233-44. doi: 10.1128/AAC.00675-10. Epub 2011 Mar 7. PMID 21383099
- [Background] Mzayek F, Deng H, Mather FJ, Wasilevich EC, Liu H, Hadi CM, Chansolme DH, Murphy HA, Melek BH, Tenaglia AN, Mushatt DM, Dreisbach AW, Lertora JJ, Krogstad DJ. Randomized dose-ranging controlled trial of AQ-13, a candidate antimalarial, and chloroquine in healthy volunteers. PLoS Clin Trials. 2007 Jan 5;2(1):e6. doi: 10.1371/journal.pctr.0020006. PMID 17213921
- [Background] Lakshmanan V, Bray PG, Verdier-Pinard D, Johnson DJ, Horrocks P, Muhle RA, Alakpa GE, Hughes RH, Ward SA, Krogstad DJ, Sidhu AB, Fidock DA. A critical role for PfCRT K76T in Plasmodium falciparum verapamil-reversible chloroquine resistance. EMBO J. 2005 Jul 6;24(13):2294-305. doi: 10.1038/sj.emboj.7600681. Epub 2005 Jun 9. PMID 15944738
- [Result] Koita OA, Sangare L, Miller HD, Sissako A, Coulibaly M, Thompson TA, Fongoro S, Diarra Y, Ba M, Maiga A, Diallo B, Mushatt DM, Mather FJ, Shaffer JG, Anwar AH, Krogstad DJ. AQ-13, an investigational antimalarial, versus artemether plus lumefantrine for the treatment of uncomplicated Plasmodium falciparum malaria: a randomised, phase 2, non-inferiority clinical trial. Lancet Infect Dis. 2017 Dec;17(12):1266-1275. doi: 10.1016/S1473-3099(17)30365-1. Epub 2017 Sep 12. PMID 28916443

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | AQ-13 | Coartem Treatment
Started | 33 | 33
Completed | 28 | 33
Not Completed | 5 | 0
Not completed — Withdrawal by Subject | 2 | 0
Not completed — Lost to Follow-up | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | AQ-13 | Coartem Treatment | Total
Number analyzed (Participants) | 33 | 33 | 66
Age, Continuous [Mean (Standard Deviation); unit: Years] | 30.3 (12.2) | 31.9 (14.8) | 31.1 (13.56)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Males | 33 | 33 | 66
Region of Enrollment [Number; unit: participants]
  Mali | 33 | 33 | 66
Haemoglobin concentration [Mean (Standard Deviation); unit: g/dL] | 12.1 (1.8) | 12.5 (2.1) | 12.3 (1.96)
Height [Mean (Standard Deviation); unit: cm] | 174.3 (7.2) | 175.5 (7.1) | 174.9 (7.15)
Weight [Mean (Standard Deviation); unit: kg] | 64.2 (7.8) | 67.5 (11.7) | 65.85 (9.94)
Median number of asexual parasites per μL [Median (Standard Deviation); unit: Asexual parasites per microliter] | 11850 (28900) | 12000 (21575) | 11925 (25501.87)
CVIET genotype parasites [Count of Participants; unit: Participants] — CVIET is the Plasmodium falciparum chloroquine resistance transporter (pfcrt) haplotypes at aminoacids 72-76
  Participants | 16 | 13 | 29
CVMNK genotype parasites [Count of Participants; unit: Participants] — CVMNK is the Plasmodium falciparum chloroquine resistance transporter (pfcrt) haplotypes at aminoacids 72-76
  Participants | 12 | 14 | 26
CVIET and CVMNK genotype parasites [Count of Participants; unit: Participants] — CVIET and CVMNK are the Plasmodium falciparum chloroquine resistance transporter (pfcrt) haplotypes at aminoacids 72-76
  Participants | 5 | 6 | 11

OUTCOME MEASURES:

1. Primary Outcome: Cure Rates of AQ-13 and Coartem for Uncomplicated Plasmodium Falciparum Malaria in Adult Malian Males.
Description: Cure rate is defined as a lack of recrudescence within 42 days PCR-corrected (correcting for new infections due to treatment failures). The investigators were looking for no evidence of recurrent infection with the same parasite genotype after reduction of the asexual parasitemia to less than 25% of the admission value by day 3 and clearance of asexual parasites and fever by day 7 to measure the cure rate. Failure is defined as lack of cure.
Time Frame: Subjects are followed for 42 days after beginning treatment with either AQ-13 or Coartem..
Measure: Count of Participants; unit: Participants
Arm/Group | AQ-13 | Coartem Treatment
Number analyzed (Participants) | 33 | 33
Participants | 28 | 31

2. Secondary Outcome: Number of Participants With Adverse Events
Description: Adverse events (AEs) are defined as events possibly related to the study drug(s) as judged by blinded physician observers that occur within 4 weeks of beginning treatment with AQ-13 or Coartem. The investigators asked participants to report the less serious adverse events (≤ grade 1) and the grade 2-4 adverse events and counted the number of participants who had those adverse events happen.
Time Frame: Within 4 weeks of beginning treatment with either AQ-13 or Coartem
Measure: Count of Participants; unit: Participants
Arm/Group | AQ-13 | Coartem Treatment
Number analyzed (Participants) | 33 | 33
Participants
  Less serious adverse events (≤ grade 1) | 32 | 33
  Grade 2-4 adverse events | 0 | 0

3. Secondary Outcome: Parasite Clearance Time
Description: Blood smears are performed at the time of diagnosis and then (for persons who have been enrolled after providing their informed consent to participate) twice daily until two successive negative smears have been obtained.
Time Frame: From the time of beginning treatment with either AQ-13 or Coartem to the first of 2 successive negative blood smears, assessed during the 1 week inpatient stay.
Measure: Mean (95% Confidence Interval); unit: Hour
Arm/Group | AQ-13 | Coartem Treatment
Number analyzed (Participants) | 33 | 33
Hour | 47.3 [43.5 to 51.1] | 32.5 [28.0 to 37.0]

4. Secondary Outcome: Number of Participants With Recrudescence of Infection
Description: Recrudescence of infection with malaria is the reactivation of the disease after treatment due to incomplete eradication of the parasite, Plasmodium. The parasites causing these recurrences had the same molecular markers as the original infections in these participants, they were considered recrudescences (late treatment failures) rather than new infections. The investigators counted the number of participants who had recrudescence of infection.
Time Frame: Within 42 days after beginning treatment with either AQ-13 or Coartem
Population: Two participants who withdrew on day 4 and three who were lost to follow-up were not included in this analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | AQ-13 | Coartem Treatment
Number analyzed (Participants) | 28 | 33
Participants | 0 | 2

5. Secondary Outcome: QTc Interval Response Following Antimalarial Treatment
Description: Corrected QT (QTc) interval was measured at antimalarial dosing and at 4 hours after dosing using HolterCare (version 10.6.0) monitors.
Time Frame: Between dosing and 4 hours after dosing
Measure: Mean (95% Confidence Interval); unit: ms
Arm/Group | AQ-13 | Coartem Treatment
Number analyzed (Participants) | 33 | 33
ms | -1.2 [-2.9 to 0] | 0.4 [-0.4 to 1.0]

6. Secondary Outcome: Mean Fever Clearance Time in Days
Description: Body temperature was measured twice daily with an electronic (digital) thermometer during the 5-7 day inpatient stay. Fever clearance time was defined as the first persistently normal temperature (<37·5°C) during week 1 of inpatient stay.
Time Frame: Days 1-7 after beginning treatment with either AQ-13 or Coartem
Measure: Mean (95% Confidence Interval); unit: Days
Arm/Group | AQ-13 | Coartem Treatment
Number analyzed (Participants) | 33 | 33
Days | 1.0 [1.0 to 1.0] | 1.23 [1.08 to 1.38]

7. Secondary Outcome: Peak Cmax
Description: One of the pharmacokinetic parameters for AQ-13 that was measured was Peak Cmax (Cmax=maximal concentration) which was calculated based on serial blood levels (35 blood level determinations of AQ-13 and its metabolites over the 42 day study period) and urine collections (24 hour collections for the first four days after beginning treatment).
Time Frame: 42 Days
Measure: Mean (95% Confidence Interval); unit: μM
Arm/Group | AQ-13
Number analyzed (Participants) | 17
μM | 2.526 [2.16 to 2.89]

8. Secondary Outcome: Time to Peak Tmax
Description: One of the pharmacokinetic parameters for AQ-13 that was measured was time to peak tmax (tmax is time from beginning treatment to the maximal concentration), which was calculated based on serial blood levels (35 blood level determinations of AQ-13 and its metabolites over the 42 day study period) and urine collections (24 hour collections for the first four days after beginning treatment).
Time Frame: 42 days
Measure: Mean (95% Confidence Interval); unit: Hours
Arm/Group | AQ-13
Number analyzed (Participants) | 17
Hours | 28.1 [27.3 to 28.9]

9. Secondary Outcome: 1-week AUC
Description: One of the pharmacokinetic parameters for AQ-13 that was measured was 1-week area under the curve (AUC) for the first 7 days, which was calculated based on serial blood levels (35 blood level determinations of AQ-13 and its metabolites over the 42 day study period) and urine collections (24 hour collections for the first four days after beginning treatment).
Time Frame: 42 days
Measure: Mean (95% Confidence Interval); unit: μM/h
Arm/Group | AQ-13
Number analyzed (Participants) | 17
μM/h | 205.4 [176.9 to 233.9]

10. Secondary Outcome: Mean Residence Time
Description: One of the pharmacokinetic parameters for AQ-13 that was measured was Mean Residence Time (MRT), which was calculated based on serial blood levels (35 blood level determinations of AQ-13 and its metabolites over the 42 day study period) and urine collections (24 hour collections for the first four days after beginning treatment).
Time Frame: 42 Days
Measure: Mean (95% Confidence Interval); unit: Days
Arm/Group | AQ-13
Number analyzed (Participants) | 17
Days | 7.19 [5.20 to 9.18]

11. Secondary Outcome: Clearance
Description: One of the pharmacokinetic parameters for AQ-13 that was measured was clearance (Cl/f), which was calculated based on serial blood levels (35 blood level determinations of AQ-13 and its metabolites over the 42 day study period) and urine collections (24 hour collections for the first four days after beginning treatment).
Time Frame: 42 Days
Measure: Mean (95% Confidence Interval); unit: L/h
Arm/Group | AQ-13
Number analyzed (Participants) | 17
L/h | 5.86 [4.81 to 6.91]

12. Secondary Outcome: Elimination t½
Description: One of the pharmacokinetic parameters for AQ-13 that was measured was elimination t½ (t½=elimination half-life) which was calculated based on serial blood levels (35 blood level determinations of AQ-13 and its metabolites over the 42 day study period) and urine collections (24 hour collections for the first four days after beginning treatment).
Time Frame: 42 Days
Measure: Mean (95% Confidence Interval); unit: Days
Arm/Group | AQ-13
Number analyzed (Participants) | 17
Days | 3.85 [2.44 to 5.26]

ADVERSE EVENTS:
Time Frame: 42 days
Arm/Group | AQ-13 | Coartem Treatment
All-Cause Mortality (participants affected / at risk) | 0/33 | 0/33
Serious Adverse Events (participants affected / at risk) | 0/33 | 0/33
Other Adverse Events (participants affected / at risk) | 32/33 | 33/33
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | AQ-13 (N=33) | Coartem Treatment (N=33)
Fever (Infections and infestations) | 32 | 29
Weakness (Musculoskeletal and connective tissue disorders) | 27 | 28
Myalgias and arthralgias (Musculoskeletal and connective tissue disorders) | 27 | 25
Headache (Nervous system disorders) | 32 | 31
Anorexia (Gastrointestinal disorders) | 24 | 20
Nausea (Gastrointestinal disorders) | 17 | 13
Vomiting (Gastrointestinal disorders) | 12 | 7
Abdominal pain (Gastrointestinal disorders) | 9 | 8
Diarrhoea (Gastrointestinal disorders) | 1 | 6
Cough (Respiratory, thoracic and mediastinal disorders) | 7 | 8
Pruritus (Skin and subcutaneous tissue disorders) | 16 | 9
Tinnitus (Ear and labyrinth disorders) | 5 | 2
Influenza-like syndrome (Respiratory, thoracic and mediastinal disorders) | 9 | 11
Temperature (Blood and lymphatic system disorders) | 16 | 13
Pallor (Gastrointestinal disorders) | 3 | 2
Jaundice (Gastrointestinal disorders) | 2 | 2

LIMITATIONS AND CAVEATS:
The Principal Investigator, Dr. Donald Krogstad, died on August 14, 2020 (see https://www.ncbi.nlm.nih.gov/pmc/articles/PMC7543845/). The Results Point of Contact has been updated to list Jeffrey G. Shaffer, PhD.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-02-13): https://cdn.clinicaltrials.gov/large-docs/64/NCT01614964/Prot_SAP_000.pdf